CLINICAL TRIAL: NCT04791527
Title: Assessing the Feasibility and Acceptability of a 12-week Online Stress Reduction/Wellness Intervention for Primary Biliary Cholangitis: a Pre-post Single-arm Interventional Study
Brief Title: Online Wellness Intervention for Primary Biliary Cholangitis (PBC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106526
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Mind Body Therapy; Stress; Quality of Life; Wellbeing; Yoga; Meditation; Psychological
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Mind-Body Therapies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-body Intervention arm (Experimental): Online yoga, meditation, behavior change tips, and nutrition tips
  Interventions: Behavioral: Mind-body therapy

INTERVENTIONS:
Behavioral: Mind-body therapy — Online yoga, meditation, behavior change tips, and nutrition tips

SUMMARY:
Primary biliary cholangitis (PBC) is a chronic autoimmune condition of the liver. Persons with PBC have high rates of liver disease-related symptoms and poor health-related quality of life - amongst the lowest of all chronic liver diseases. Patients and the Canadian PBC Society have identified the need for self-care tools to manage symptom burden. Building upon a previously developed online wellness program for inflammatory bowel disease (IBD), the researchers have developed a mind-body wellness module specific for patients with PBC. The 12 week module will be delivered online, and each week is made of an introduction video, 15-20 minutes of yoga, 10-15 minutes of meditation, behavior change tips, and nutrition tips. In a pre-post single arm feasibility study, the researchers will assess how acceptable this module is to patients through looking at rates of refusal, completion rates, and patient feedback. At the beginning and the end of the 12-week research study, participants will complete surveys to assess exploratory outcome measures including stress, anxiety, depression, resilience, quality of life, fatigue, and perceived ability to participate in the 12 week module. After the program, the research team will conduct interviews with participants to allow them to share their other feedback about the program. The researchers will also send surveys to the participants one month after the program ends to asses their continued satisfaction with and adherence to the program.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Identified diagnosis of PBC
* HADS score <=10
* English language proficiency to complete questionnaires and read the educational material
* Access to the Internet and a computer or smart device at home.

Exclusion Criteria:

* Patients with a major medical co-morbidity
* Inability to provide informed written consent
* Severe psychiatric disorders (HADS scores >10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 12 Weeks
  The degree to which situations in one's life are appraised as stressful will be assessed using the Perceived Stress Scale. The minimum score is 0, the maximum score is 40, and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
HADS Anxiety and Depression Scale | 12 Weeks
  Depression and anxiety will be measured on the Hospital Anxiety and Depression Scale. The minimum value is 0, the maximum is 21, and higher scores mean a worse outcome.
PBC-40 | 12 Weeks
  Six PBC specific quality of life domains will be measured on the PBC-40. For each question, the minimum value is 1, the maximum value is 5, and 5 indicates a worse outcome. The overall scoring range varies among domains.
Modified Fatigue Impact Scale | 12 Weeks
  The effect of fatigue on cognitive, physical, and psychosocial functioning will be measured with the modified fatigue impact scale. The minimum value is 0, the maximum value is 36, and higher scores mean a worse outcome.
Connor Davidson Resilience Scale 10 | 12 Weeks
  Resilience will be measured on the Connor Davidson Resilience Scale 10. The minimum value is 0, the maximum value is 40, and higher scores indicate a better outcome.
Capability, Opportunity, Motivation, Behavior (COM-B) Survey | 12 Weeks
  Capability, opportunity, and motivation for behavior change will be measured on the COM-B survey. The lowest score is 0, the highest score is 60, and higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Puneeta Tandon, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Watt M, Spence JC, Tandon P. Development of a Theoretically Informed Web-Based Mind-Body Wellness Intervention for Patients With Primary Biliary Cholangitis: Formative Study. JMIR Form Res. 2021 Oct 8;5(10):e29064. doi: 10.2196/29064. PMID 34623317